CLINICAL TRIAL: NCT02410525
Title: A Phase 1, Open-label, 3-period, Randomized, Partially Fixed Sequence, 2-way Crossover Study With A Microdose Of [11c]Pf-06427878 Administered With And Without Two Non-radioactive Doses Of Pf-06427878 To Characterize Tissue Distribution Using Positron Emission Tomography In Healthy Adult Male Subjects
Brief Title: A Study Testing A Radioactive Compound Given Through A Vein With And Without The Non-Radioactive Compound, Given By Mouth, To Characterize Tissue Distribution Using Positron Emission Tomography Scanning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7871003
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: hyperlipidemia; positron emission tomography
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- [11C]PF-06427878 (Experimental): Single intravenous infusion of [11C]PF-06427878 in Periods 1, 2 and 3 to investigate the liver and plasma radioactivity, radioactivity in organs relative to plasma, pharmacokinetics, and safety and tolerability
  Interventions: Drug: [11C]PF-06427878
- PF-06427878 10 mg (Experimental): Single oral dose of 10 mg PF-06427878 in Period 2 or 3 to investigate the liver and plasma radioactivity, radioactivity in organs relative to plasma, pharmacokinetics, and safety and tolerability
  Interventions: Drug: PF-06427878 10 mg
- PF-06427878 600 mg (Experimental): Single oral dose of 600 mg PF-06427878 in Period 2 or 3 to investigate the liver and plasma radioactivity, radioactivity in organs relative to plasma, pharmacokinetics, and safety and tolerability
  Interventions: Drug: PF-06427878 600 mg

INTERVENTIONS:
Drug: [11C]PF-06427878 — Single administration via intravenous infusion of 20 ug [11C]PF-06427878 on Day 1 of all 3 Periods
  Arms: [11C]PF-06427878
Drug: PF-06427878 10 mg — Single oral administration of 10 mg PF-06427878 on Day 1 of Period 2 or 3, at approximately 2.5 hours prior to [11C]PF-06427878 administration
  Arms: PF-06427878 10 mg
Drug: PF-06427878 600 mg — Single oral administration of 600 mg PF-06427878 on Day 1 of Period 2 or 3, at approximately 2.5 hours prior to [11C]PF-06427878 administration
  Arms: PF-06427878 600 mg

SUMMARY:
In this study, radioactive PF-06427878 will be administered, through a vein, alone and with 2 different oral doses of non-radioactive PF-06427878 to healthy, adult, male subjects. Positron emission tomography will be used to characterize tissue distribution. The study will also characterize how the study drug behaves in the body, its safety, and how the body tolerates it.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* body mass index 17.5-30.5 kg/m2 ; body weight >50 kg
* signed and dated informed consent document
* willing and able to comply with study requirements

Exclusion Criteria:

* tobacco/nicotine containing products > equivalent of 5 cigarettes per day
* history of cumulative ionizing radiation exposure in the past year, including anticipated exposure in this study, and subjects with current, past or anticipated exposure to radiation in the workplace
* severe claustrophobia
* unable to lie still for the required period to acquire images

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percent injected radioactivity (per gram) over time in the liver | All Periods;Day 1;0-120min
Percent injected radioactivity (per gram) over time in the plasma | All Periods;Day 1;0hr,1,2,3,4,5,5.5,6,6.5,7,8,9,10,12,15,20,25,30,40,50,60,75,90,105,120min

SECONDARY OUTCOMES:
Relative radioactivity in liver versus plasma | All Periods;Day 1;0hr,1,2,3,4,5,5.5,6,6.5,7,8,9,10,12,15,20,25,30,40,50,60,75,90,105,120min
  Ratio of AUC of percent injected radioactivity (per gram) over time in liver to AUC of percent injected radioactivity (per gram) over time in plasma
Time-course of total radioactivity as percentage of injected radioactivity (per gram) in the gall bladder, if this region is identifiable | All Periods;Day 1;0-2hr
% of parent in plasma over time | All Periods;Day 1;0hr,1,2,3,4,5,5.5,6,6.5,7,8,9,10,12,15,20,25,30,40,50,60,75,90,105,120min
  Parent is study drug PF-06427878
Plasma PK of PF-06427878: AUClast, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: AUClast, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min
Time-course of total radioactivity as percentage of injected radioactivity (per gram) in the biliary tree, if this region is identifiable | All Periods;Day 1;0-2hr
Time-course of total radioactivity as percentage of injected radioactivity (per gram) in the abdominal fat, if this region is identifiable | All Periods;Day 1;0-2hr
Time-course of total radioactivity as percentage of injected radioactivity (per gram) in the kidney, if this region is identifiable | All Periods;Day 1;0-2hr
Time-course of total radioactivity as percentage of injected radioactivity (per gram) in the urinary bladder, if this region is identifiable | All Periods;Day 1;0-2hr
Time-course of total radioactivity as percentage of injected radioactivity (per gram) in the thigh muscle, if this region is identifiable | All Periods;Day 1;0-2hr
Plasma PK of PF-06427878: AUCinf, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: Cmax, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: Tmax, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: t½, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: CL, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: Vss, as data permit | Period 1;Day 1;0,3,5,15,30,60,90,120,135min
Plasma PK of PF-06427878: Vss, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min
Plasma PK of PF-06427878: AUCinf, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min
Plasma PK of PF-06427878: Cmax, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min
Plasma PK of PF-06427878: Tmax, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min
Plasma PK of PF-06427878: t½, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min
Plasma PK of PF-06427878: CL/F, as data permit. | Periods 2 & 3;Day 1;prebreakfast,-90,-60,0,120min

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Anylan Center, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut